CLINICAL TRIAL: NCT01483014
Title: Phase ll Study of Imatinib Mesylate for the Neoadjuvant Treatment of Patients With Gastrointestinal Stromal Tumors (GIST)
Acronym: CONVERT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BBR10
Record Dates: First submitted 2011-11-29; First posted 2011-12-01 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal,; stromal,; neoadjuvant,; imatinib,; mesylate,; pre-operatory
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

ARMS (1):
- imatinib (Experimental)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
This study will evaluate the efficacy, safety, tolerability of imatinib in the neoadjuvant treatment (pre-operatory) of patients with GIST. It will also evaluate the potential of imatinib to convert a tumor from inoperable to operable.

ELIGIBILITY:
Inclusion Criteria:

* patients with age between 18 and 80 years
* diagnosis of GIST not previously treated
* Patients will be included in the protocol regardless of operability; in the case of an operable tumor, patients are eligible if, in the opinion of the surgeon, resection would be suboptimal, disfiguring or functionally disabling (i.e. incomplete resection or other which cold compromise severely the quality of life or other GI function)

Exclusion criteria:

* presence of metastatic disease
* use of other antineoplastic treatment (chemotherapy, immunotherapy, radiotherapy)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Objective response using the RECIST criteria | 16 weeks

SECONDARY OUTCOMES:
Progression free survival | 16 weeks
Time and duration of response | 16 weeks
Time to treatment failure | 16 weeks
Overall survival | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Brazil (9):
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investivative site, Belo Horizonte
  - Novartis Investivative site, Florianópolis
  - Novartis Investivative site, Porto Alegre
  - Novartis Investivative site, Rio de Janeiro
  - Novartis Investivative site, São Paulo